CLINICAL TRIAL: NCT05169073
Title: The Impact of 3D Virtual Reality MRCP Rendering on Surgical Performance During Laparoscopic Cholecystectomy: A Pilot Study
Brief Title: Virtual Reality Training for Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CU621
Record Dates: First submitted 2021-12-07; First posted 2021-12-23 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Virtual Reality; Gallbladder; Bile Duct Injury; Medical Education; Laparoscopy

STUDY DESIGN:
Intervention Model Description: The order in which the operations will be performed by each resident is random.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor and analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality MRCP (Experimental): The MRCP images will be transferred into a 3D VR rendering software (Specto VR TM) for each patient. Residents will have the opportunity to use the virtual reality environment the day before surgery until a sufficient understanding of the anatomy is achieved.
  Interventions: Procedure: Virtual Reality training
- Conventional MRCP (Active Comparator): Controls will have regular access to the conventional MRCP images.
  Interventions: Procedure: Conventional training

INTERVENTIONS:
Procedure: Virtual Reality training — In the Virtual Reality (VR) study arm, a VR software (Specto VRTM, version 4.0, Diffuse Ltd, Heimberg, Switzerland) will be used to display volumetric MRCP data using a tethered head-mounted display (HMD) prior to the operation. Specto uses volume rendering at 180 frames/sec to visualize the medical data in an immersive fashion in the VR environment and allows for viewing of the 3D reconstructed 3D imaging with 360° free movement. Each participant will perform a procedure with VR training and one with conventional preparation (MRCP).
  Arms: Virtual Reality MRCP
Procedure: Conventional training — In the conventional study arm, the participants will view the preoperative MRCP.
  Arms: Conventional MRCP

SUMMARY:
Cholecystectomy is one the most frequent laparoscopic procedures worldwide. It is a safe and effective operation but intraoperative bile duct injury remains a relevant complication with serious consequences for the patient. Most of the complications occur due to a lack of knowledge of the anatomy or misidentification of the cystic duct. Thus, the study of the anatomy is a cornerstone of a successful procedure and the preoperative magnetic resonance cholangiopancreatography (MRCP) is a way to preoperatively determine relevant structures to avoid intraoperative incidents.

This trial has been designed to assess the effect of preoperative virtual reality training based on MRCP on intraoperative performance and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Referred for elective cholecystectomy for symptomatic cholecystolithiasis/chronic cholecystitis
* Early cholecystectomy after acute biliary pancreatitis
* Concomitant minor procedures (adhesiolysis, umbilical hernia repair, liver biopsy)
* Sufficient quality of MRCP

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) classification ≥ 4
* Previous major open upper abdominal surgery
* Suspicion for concomitant biliary disease (e.g. Mirizzi-Syndrome)
* Robotic cholecystectomy
* Planned open procedures

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Global Assessment of Laparoscopic Skills (GOALS) score assessed by assisting surgeon | On the day of surgery (within 12 hours)
  For the global assessment of laparoscopic skills, the Global Operative Assessment of Laparoscopic Skills (GOALS) will be used. Evaluation will be performed by the attending surgeon. The GOALS is a 5 item rating scale and the items are scored using a 5-point Likert scale where "1" represents the lowest level of performance, and "5" is considered ideal performance. The total score for the global rating scale is the sum of the scores for each of the 5 items for a maximum total score of 25.

SECONDARY OUTCOMES:
Global Assessment of Laparoscopic Skills (GOALS) score assessed by resident | On the day of surgery (within 12 hours)
  For the global assessment of laparoscopic skills, the Global Operative Assessment of Laparoscopic Skills (GOALS) will be used. Evaluation will be performed by the resident (self-assessment).
Critical View of Safety | Postoperative within 30 days (Video-Analysis)
  The "Sanford-Strasberg' Critical-view-of-safety (CVS)" is a method for judging the CVS objectively through intraoperative photographs. It evaluates the CVS captured by anterior and posterior ("doublet") views. The minimum score is 0, and the maximum is 6. The higher the score, the more satisfactory is the CVS. The "Sanford-Strasberg' CVS Score" is useful in evaluating the CVS in video records and the CVS has been recognized as an essential and effective security method to reduce the risk of bile duct injury.
Time to critical view of safety | Postoperative within 30 days (Video-Analysis)
  Time required to achieve the CVS or i.e. until the clips are placed during the operation.
Efficiency improvement | On the day of surgery (within 12 hours)
  Discrepancy between actual and planned operative time
Self-confidence | On the day of surgery (within 12 hours)
  The self-confidence scale is a psychometrically valid tool to measure residents' self-confidence during surgical learning. Self-rating will be performed by selection of 6 items, each on a Likert scale ranging from 1 to 5. The maximum score attainable is 30 and the higher the score, the higher the self-confidence.
Operative time | During surgery
  Time from incision to wound closure
Intraoperative interventions by assisting surgeon | During surgery
  Any intervention necessary to guide to resident. I.e. whenever the assisting surgeon takes over the position of the operating surgeon.

OTHER OUTCOMES:
Length of hospital stay | At the day of discharge
  Length of the total hospital stay (days)
90-day postoperative Complications | Until 90 days after surgery
  All postoperative deviations from the normal expected course graded according to the Accordion classification and the comprehensive complication index.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Staubli, MD, Principal Investigator — Clarunis - University Center for Gastrointestinal and Liver Diseases
Locations (1):
- University Centre for Gastrointesintal and Liver Disease, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nassar AHM, Ashkar KA, Mohamed AY, Hafiz AA. Is laparoscopic cholecystectomy possible without video technology? Minimally Invasive Therapy. 1995; 4:2 63-65
- [Background] Vassiliou MC, Feldman LS, Andrew CG, Bergman S, Leffondre K, Stanbridge D, Fried GM. A global assessment tool for evaluation of intraoperative laparoscopic skills. Am J Surg. 2005 Jul;190(1):107-13. doi: 10.1016/j.amjsurg.2005.04.004. PMID 15972181
- [Background] Sanford DE, Strasberg SM. A simple effective method for generation of a permanent record of the Critical View of Safety during laparoscopic cholecystectomy by intraoperative "doublet" photography. J Am Coll Surg. 2014 Feb;218(2):170-8. doi: 10.1016/j.jamcollsurg.2013.11.003. Epub 2013 Nov 9. PMID 24440064
- [Background] Geoffrion R, Lee T, Singer J. Validating a self-confidence scale for surgical trainees. J Obstet Gynaecol Can. 2013 Apr;35(4):355-361. doi: 10.1016/S1701-2163(15)30964-6. PMID 23660044